CLINICAL TRIAL: NCT05545254
Title: Health-promoting Lifestyle of Breast Cancer Patients and Family Members in a Chinese Genetic Counseling Clinic: A Cross-sectional Study
Brief Title: Health-promoting Lifestyle in a Genetic Counseling Clinic
Status: Completed | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhenqi Lu, Director of nursing department, Fudan University
Other Study IDs: FNF201830
Record Dates: First submitted 2022-09-09; First posted 2022-09-19 (Actual); Last update posted 2022-09-19 (Actual); Status verified 2022-09

CONDITIONS: Breast Cancer; Genetic Testing
Keywords: Health-promoting lifestyle, breast cancer, genetic
MeSH Terms: conditions — Breast Neoplasms | interventions — Genetic Testing

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Breast cancer patients and their family members who have undertaken genetic testing: In this study, 259 participants were recruited from November 2019 to March 2022. All participants originated from a genetic counseling clinic of a cancer center in Shanghai, China. 259 participants were contact, and among them, 158 participants finally agreed to participate and completed the survey.
  Interventions: Genetic: genetic testing

INTERVENTIONS:
Genetic: genetic testing — Two questionnaires were included in the link, one referring to the demographic information, and another one involving the health-promoting lifestyle. In the demographic information, the genetic test results were not requested to be written, but the participants need to answer whether they understand the results. The HPLP-Ⅱ is an scale instrument used to evaluate a person's health-promoting lifestyle behaviors, which contains 52 items and has been translated into Chinese in 1997. It contains 6 subscales: self-actualization, health responsibility, physical activity, nutrition, interpersonal relationships and stress management.

SUMMARY:
This was a cross-seThis was a cross-sectional study, which aimed to describe the health-promoting lifestyle of breast cancer patients and family members in a Chinese genetic counseling clinic, and to explore its various levels with different socio-economic variables. 259 patients conformed to the inclusion and exclusion criteria were enrolled. Participants were sent a questionnaire web-link to be invited to finish this survey. 140 participants were finally included in this study. Finally, a good level of health-promoting lifestyle of breast cancer patients and family members was acquired. More education and intervention should be tailored to enhance and encourage health-promoting lifestyle behaviors in participants with low monthly family income. Additionally, developing nutritional curriculum and strengthening the publicity of nutritional popular science were priorities in the future improvement measures.ctional study

DETAILED DESCRIPTION:
Purpose: This study aimed to describe the health-promoting lifestyle of breast cancer patients and family members in a Chinese genetic counseling clinic, and to explore its various levels with different socio-economic variables.

Method: This was a cross-sectional study. The participants in this study originated from a genetic counseling clinic of a cancer center in Shanghai, China. 259 patients conformed to the inclusion and exclusion criteria were screened and contact from November 2019 to March 2022. Participants agreed to participate were sent a questionnaire web-link to be invited to finish this survey. Two questionnaires were included in the link, one referring to the socio-economic information, the other referring to the health-promoting lifestyle. Chinese Health-promoting lifestyle profile-Ⅱ(HPLP-Ⅱ) was used to evaluate the health-promoting lifestyle.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years old;
* with a diagnosis of breast cancer or having a family history of breast cancer
* the first time to take genetic testing in our clinic
* ECOG<2.

Exclusion Criteria:

* diagnosed with psychiatric or intellectual impairment
* having a history of genetic testing previously

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: In this study, 259 participants were recruited from November 2019 to March 2022. All participants originated from a genetic counseling clinic of a cancer center in Shanghai, China. 259 participants were contact, and among them, 158 participants finally agreed to participate and completed the survey.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2019-11-13 (Actual); Primary Completion 2022-03-04 (Actual); Study Completion 2022-03-04 (Actual)

PRIMARY OUTCOMES:
Chinese Health-promoting lifestyle profile-Ⅱ | The primary outcome was measured during one month after the genetic test.
  HPLP-Ⅱ is an scale instrument used to evaluate a person's health-promoting lifestyle behaviors, which contains 52 items and has been translated into Chinese in 1997.It contains 6 subscales: self-actualization, health responsibility, physical activity, nutrition, interpersonal relationships and stress management. A Likert 4-scale is used to measure each item, and never to regularly signifies 1-4. The total score ranges from 52 to 208. Higher scores mean better health-promoting behaviors.

CONTACTS AND LOCATIONS:
Overall Officials: Zhenqi Lu, Master, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: No